CLINICAL TRIAL: NCT04598204
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of Rapamycin in Complex Vascular Anomalies in Pediatric Patients
Brief Title: Efficacy and Safety of Rapamycin to Complex Vascular Anomalies in Pediatric Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-EKZX-003
Record Dates: First submitted 2020-06-28; First posted 2020-10-22 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Vascular Anomalies
Keywords: Rapamycin
MeSH Terms: conditions — Vascular Malformations | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): To treat the enrolled patients with oral rapamycin at an initial dosage of 0.8mg/m2, once daily for children under 3 years old and twice daily (every 12 hours) for those above 3 years, and adjust the dosage to target a trough concentration of rapamycin in plasma as 10-15ng/ml （OR 15-20ng/ml if the efficacy of treatment is not satisfactory）. One course lasts for 12weeks and no more than 4 course is given.
  Interventions: Drug: Treatment with oral rapmycin

INTERVENTIONS:
Drug: Treatment with oral rapmycin — To treat the enrolled patients with oral rapamycin with an initial dosage of 0.8mg/m2, once daily for children under 3 years old and twice daily (every 12 hours) for those above 3 years, and adjust the dosage to target a trough concentration of rapamycin in plasma as 10-15ng/ml （OR 15-20ng/ml if the efficacy of treatment is not satisfactory）. One course lasts for 12weeks and no more than 4 course is given.

SUMMARY:
KHE and TA are rare tumors and some of the cases may lead to life-threatening complications including Kasabach-Merritt Phenomenon. Typically treated with steroids and vincristine, a majority of the cases do not have good prognosis. Complex vascular malformations are always managed by surgery,sclerotherapy and embolization therapy. While many of the cases still lead to complications such as disfigurement, chronic pain, recurrent infections, coagulopathies. Different medical centers are exploring new therapy for these tough problems. This study is plotted to determine the efficacy and safety of rapamycin monotherapy in KHE/TA and complex vascular malformations in pediatric patients.

DETAILED DESCRIPTION:
According to the classification （revised in 2014）by International Society for the Study of Vascular （ISSVA ）, vascular anomalies are classified into two distinct disease entities，including vascular tumors and vascular malformations differing in their biologic and pathologic features. Vascular tumors include infantile and congenital hemangiomas, Tufted angiomas (TA), and Kaposiform hemangioendotheliomas (KHE). Vascular malformations are classified according to their vascular tissue of origin which include capillary, venous, arteriovenous, lymphatic, and mixed malformations. Infantile hemangiomas, the most common vascular anomaly, generally have a good prognosis due to its specific biological characteristics（a predetermined life cycle from proliferation to subsequent involution). However，KHE and TA are rare vascular tumors with incidence less than 1/1000000 and along with complex lymphatic malformations and complex mixed malformations，are difficult to be successfully treated resulting in clinical problems such as disfigurement, chronic pain, recurrent infections, coagulopathies (thrombotic and hemorrhagic,including life-threatening Kasabach-Merritt Phenomenon), organ dysfunction. Rapamycin directly inhibits the mTOR pathway, thereby inhibiting cell proliferation and angio/lymphangiogenesis and is recently applied to refractory vascular . Preclinical data and case reports have confirm that rapamycin is effective for KHE/TA and some slow-flow vascular malformations. The overall goal of this trial is to objectively determine the effectiveness and safety of rapamycin monotherapy in KHE/TA and complex vascular malformations in pediatric patients and to explore the rational doses. In this study, 30 patients (aged from 1 month to 14 years old) diagnosed with KHE/TA or complex vascular that respond poorly to propranolol hydrochloride and corticosteroid are enrolled. Oral rapamycin is given as a monotherapy at a initial dose of 0.8mg/m2, once daily for children under 3 years old and twice daily (every 12 hours) for those above 3 years. And further dosage is adjusted to target a trough concentration of rapamycin in plasma as 10-15ng/ml （OR 15-20ng/ml if the efficacy of treatment is not satisfactory with concentration at 10-15ng/ml. One course lasts for 12weeks and no more than 4 courses are given.Volumetric changes as the primary outcome measure will be analysed by magnetic resonance imaging (MRI) and/or ultrasonography. Frequency of adverse events as assessed by CTCAE v4.0 is calculated to evaluate the safety of rapamycin.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: All patients must be diagnosed with Kaposiform Hemangioendotheliomas ，Tufted Angioma or complicated vascular malformation as determined by clinical, radiographic and histologic criteria (when possible)；
2. Patients must have vascular anomalies that respond poorly to propranolol hydrochloride and corticosteroid;
3. Organ function requirements:

   3.1 Adequate liver function defined as: Total bilirubin (sum of conjugated and unconjugated) ≤1.5 x ULN for age, and SGPT (ALT) <5 x ULN for age, and Serum albumin > or = 2 g/dL.

   3.2 Adequate Bone Marrow Function defined as: Peripheral absolute neutrophil count (ANC) > or = 1000/microL Hemoglobin > or = 8.0 gm/dL (may receive RBC transfusions) Platelet count > or = 50,000/microL (transfusion independent defined as not receiving a platelet transfusion within a 7 day period prior to enrollment) （Note: There is NO platelet requirement for patients with Kasabach-Merritt Phenomenon） 3.3 Adequate Renal Function Defined as:

   A serum creatinine based on age as follows:

   ≤ 5 years of age maximum serum creatinine (mg/dL) of 0.8 6 < age ≤ 10 years of age maximum serum creatinine (mg/dL) of 1.0 11 < age ≤ 15 years of age maximum serum creatinine (mg/dL) of 1.2 > 15 years of age maximum serum creatinine (mg/dL) of 1.5 cystatin C equal to or less than the upper limit of normal for the patient. If cystatin C does not initially meet this criterion, it may be repeated or a more sensitive screening by nuclear GFR must be ≥ 70 ml/min.

   Urine protein to creatinine ratio (UPC) < 0.3 g/l
4. Patients must be Human Immunodeficiency Virus negative and without immunodeficiency or infectious disease such as viral hepatitis.
5. Patients must have no gastrointestinal disease that would affect the absorption of rapamycin.
6. Performance Status: Karnofsky > or = 50 (>10 years of age) and Lansky > or = 50 for patients < or = 10 years of age.
7. Patients may not be currently receiving strong inhibitors of CYP3A4 or strong inducers of CYP3A4 and may not have received these medications within 1 week of entry.
8. Patients must not have corticosteroid, chemotherapy or radiotherapy within 2 weeks of entry.
9. Guardians must be informed consent.

Exclusion Criteria:

1. Known allergy to mTOR inhibitor
2. Under the treatment of other medicine for vascular anomalies.
3. Known chronic or infectious disease.
4. Patients who received prior per os treatment with an mTOR inhibitor.
5. Known digestive disease that would affect the absorption of rapamycin.
6. Guardians disagree to sign the informed consent.
7. Patients who in the opinion of the investigator would be at risk in the study or would affect the accuracy of the study results.-

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Volumetric changes in complicated vascular anomalies after rapamycin treatment | Baseline,and every 6 months until half a year after the finish of rapamycin treatment
  Response to rapamycin treatment was measured by volumetric magnetic resonance imaging (MRI) and/or ultrasonography analyses. Changes in size of vascular anomalies were classified as further growth (increase of ≥20%), no change (<20% increase and <20% decrease),and involution (decrease of ≥20%).
Time of clinical lab indexes to be improved and stable | at least weekly before a improved and stable state is reached,assessed up to 8 weeks
  For cases complicated with Kasabach-Merritt Phenomenon, clinical lab indexes including blood platelet and fibrinogen are followed up at least weekly before a improved and stable state is reached. Time (days) from the onset of treatment till these indexes to be improved and stable is calculated. Improved hematologic parameters are defined as a platelet count greater than 50,000/uL (or a 2 times increase in platelet count compared to baseline) and a fibrinogen level greater than 100mg/dl.
Occurrence of adverse reactions | From the date of trial until the date of first documented progression or date of lost to follow-up,till half a year after finish of treatment.
  Record the time, degree and outcome of adverse reactions according to Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Trough concentration of rapamycin in plasma | 5 days after the onset of rapamycin or after the adjustment of drug doses;every 3 three months during the therapy if the concentration result is in the optimal target range during the treatment,assessed up to 100 months.
  Trough concentration of rapamycin in plasma is monitored and according to which the dosage is adjusted，thus is part of the efficacy evaluation.
Evolution of clinical situation and the quality of life | Baselin,3,6,12months,and till half an year after finish of treatment
  Evolution of clinical situation and the quality of life is judged by the proxies of patients by describing clinical symptoms and by recording and viewing standardized digital photographs.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drolet BA, Trenor CC 3rd, Brandao LR, Chiu YE, Chun RH, Dasgupta R, Garzon MC, Hammill AM, Johnson CM, Tlougan B, Blei F, David M, Elluru R, Frieden IJ, Friedlander SF, Iacobas I, Jensen JN, King DM, Lee MT, Nelson S, Patel M, Pope E, Powell J, Seefeldt M, Siegel DH, Kelly M, Adams DM. Consensus-derived practice standards plan for complicated Kaposiform hemangioendothelioma. J Pediatr. 2013 Jul;163(1):285-91. doi: 10.1016/j.jpeds.2013.03.080. No abstract available. PMID 23796341